CLINICAL TRIAL: NCT02131571
Title: Prevalence of Vertebral Fractures in HIV Infected Patients Older Than 50 Years: Importance of Bone Mineral Density and Bone Biomarkers
Brief Title: Prevalence of Vertebral Fractures in HIV Infected Patients Older Than 50 Years
Acronym: FractaVIH
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: FractaVIH 117/13; EC 117/13 (Other: Ethics Committee registry)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Vertebral Fractures
Keywords: HIV; bone; fractures; vitamin D; biomarkers
MeSH Terms: conditions — Spinal Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV patients older than 50 years: HIV infected patients older than 50 years in current follow up

SUMMARY:
Prospective cohort study to determine the prevalence of vertebral fractures in HIV infected patients older than 50 years.

DETAILED DESCRIPTION:
To determine the prevalence of asymptomatic vertebral fractures in HIV patients older than 50 years, and the risk of fracture during a follow up of 2 years, according to bone mineral density at inclusion, the level of serum bone biomarkers, and the presence of secondary factors such as hypovitaminosis D or/and secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Age above 50 years
* HIV infection

Exclusion Criteria:

* Pregnancy
* Receiving corticosteroids or antiresorptive therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients older than 50 years
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of vertebral fractures in HIV patients older than 50 years | 2 years
  To determine by lumbar and thoracic x ray the presence of vertebral fractures and the changes in vertebral form or size, according to Genant methods

SECONDARY OUTCOMES:
Risk of vertebral alteration according to bone mineral density and serum biomarkers | 2 years
  To determine the relationships of vertebral alterations with bone mineral density by dual X-ray absorptiometry
Vertebral alterations during follow up | 2 years
  To determine the emergence of vertebral alterations during 2 years of follow up according to bone mineral density, bone biomarkers (osteocalcin, beta-crosslaps), and vitamin D/parathyroid hormone (PTH) status.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, MD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided